CLINICAL TRIAL: NCT06845423
Title: Prevention of Postpartum Venous Thromboembolism in Women at Intermediate Risk. An Open-label, Randomized, Controlled Trial Comparing Two Strategies With or Without Pharmacological Thromboprophylaxis
Brief Title: Prevention of Postpartum Venous Thromboembolism in Women at Intermediate Risk
Acronym: MUM-VTE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 29BRC22.0254
Record Dates: First submitted 2025-02-20; First posted 2025-02-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Venous Thromboembolism (VTE); Post Partum Women
MeSH Terms: conditions — Venous Thromboembolism | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Intervention Model Description: This is a multicenter PROBE study (prospective randomized open with blinded evaluation of the endpoints by an independent adjudication committee) with two parallel groups
Who Masked: Outcomes Assessor
Masking Description: All critical events (VTE, bleeding and mortality) will be validated by a central, independent clinical events committee (ICEC) which will adjudicate outcomes blinded for treatment allocation (PROBE study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pharmacological thromboprophylaxis using LMWH at preventive dosage. The choice of subcutaneous LMWH depends on the practice of each center:
  * Enoxaparine 4000 UI (weight > 90 kg 6000 UI)
  * Tinzaparine 3500 UI (weight > 90 kg 4500 UI)
  * Dalteparine 5000 UI (weight > 90 kg 7500 UI)
  * Nadroparine 2850 UI (weight > 90 kg 3800 UI).
  All patients can have compression stockings
  Interventions: Drug: Low molecular weight heparin
- Control group (No Intervention): No pharmacological thromboprophylaxis. All patients can have compression stockings.

INTERVENTIONS:
Drug: Low molecular weight heparin — Pharmacological thromboprophylaxis using LMWH at preventive dosage. The choice of subcutaneous LMWH depends on the practice of each center:
  * Enoxaparine 4000 UI (weight > 90 kg 6000 UI)
  * Tinzaparine 3500 UI (weight > 90 kg 4500 UI)
  * Dalteparine 5000 UI (weight > 90 kg 7500 UI)
  * Nadroparine 2850 UI (weight > 90 kg 3800 UI).
  Arms: Experimental Group

SUMMARY:
Venous thromboembolism (VTE) is currently the second cause of death in women of reproductive age worldwide. The incidence of VTE during pregnancy is 1.2 to 1.4/1000 women, half of VTE occurring during postpartum and as PE in majority of cases, accounting for 8.8% of maternal deaths.

Majority of postpartum VTE occurs in women with one or more moderate risk factors (obesity, caesarean section, postpartum hemorrhage). For these women at intermediate risk, the efficacy and safety of thromboprophylaxis have not been assessed yet during postpartum and international guidelines for pharmacological thromboprophylaxis, based on data extrapolated from other populations, observational studies and small clinical trials are inconsistent across countries.

We designed an open-label, randomized, controlled trial, aiming to demonstrate the superiority of a pharmacological thromboprophylaxis strategy with LMWH (LMWH type chosen according to physician / patient's preference) during 6 weeks after delivery (the 6-weeks follow-up visit being matched with usual care) in women at intermediate risk, over no pharmacological thromboprophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Women at intermediate risk of VTE during post-partum= with a 3% or more risk of VTE based on a validated prediction model* or International guidelines (ACCP 2012).
* Age over 18 years
* Delivery between 6 hours and < 36 hours
* Written informed consent

  * Definition: Intermediate risk is defined as ≥ 3%, based on risk prediction model developed by Sultan et al taking in account: smoking, varicose veins, obesity, comorbidities, diabetes, pre-eclampsia, post-partum hemorrhage, postpartum infection, emergency or elective section or following ACCP guidelines: one major risk factor or two minor risk factors.

Exclusion Criteria:

* Previous personal history of VTE
* LMWH started during antenatal period
* Need for anticoagulation at curative dose
* Contraindication to LMWH (previous heparin induced thrombopenia, hemostatic impairment, known severe renal insufficiency)
* Women who received more than two doses of LMWH since delivery
* Unable or refusal to give informed consent
* Aspirin at a daily dose 100 mg or dual antiplatelet therapy
* Previous inclusion in Mum-VTE study
* Concomitant participation in another therapeutic study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-05-16 (Actual); Primary Completion 2028-05-16 (Estimated); Study Completion 2028-08-16 (Estimated)

PRIMARY OUTCOMES:
Symptomatic VTE (DVT or non-fatal or fatal PE) | 6 weeks
  Blindly adjudicated objectively confirmed symptomatic VTE (DVT or non-fatal or fatal PE) ) during the first 6-week postpartum period

SECONDARY OUTCOMES:
Symptomatic VTE (DVT or non-fatal or fatal PE) | 3 months
  blindly adjudicated objectively confirmed symptomatic VTE (DVT or non-fatal or fatal PE) during 3-month follow-up period after delivery (entire study period).
Major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) | 6 weeks
  Blindly adjudicated major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) during 6-week study treatment period
Major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) | 3 months
  Blindly adjudicated major bleeding (as defined by the criteria of the International Society of Thrombosis and Haemostasis) during 3-month follow-up after delivery.
Clinically relevant non-major bleeding | 6 weeks
  Blindly adjudicated clinically relevant non-major bleeding during 6-week study treatment period
Clinically relevant non-major bleeding | 3 months
  Blindly adjudicated clinically relevant non-major bleeding during 3-month follow-up after delivery.
Net Clinical benefit | 6 weeks
  The net clinical benefit of study treatment (composite of symptomatic VTE and major or clinically relevant non major bleeding) during 6-week postpartum period
Net Clinical benefit | 3 months
  The net clinical benefit of study treatment (composite of symptomatic VTE and major or clinically relevant non major bleeding) during 3-month follow-up after delivery
Number of Thrombocytopenia | 6 weeks
  Cases of heparin induced thrombocytopenia associated with LMWH during 6-week study treatment period.
Mortality | 6 weeks
  Blindly adjudicated mortality of all causes during 6-week study treatment period
Mortality | 3 months
  Blindly adjudicated mortality of all causes during 3-month follow-up period after delivery.
VTE suspicion | 6 weeks
  Number of VTE suspicion in interventional and control arm during 6-week study treatment period
VTE suspicion | 3 months
  Number of VTE suspicion in interventional and control arm during 3-month follow-up period after delivery.
Treatment compliance | 6 weeks
  Treatment compliance during 6-week study treatment period based on Girerd questionnaire
Objectively confirmed symptomatic VTE (DVT or non-fatal or fatal PE) | 6 weeks
  - Blindly adjudicated objectively confirmed symptomatic VTE (DVT or non-fatal or fatal PE) during the first 6-week postpartum period (i.e., study treatment period) in clinically relevant prespecified subgroups (caesarean section, obesity, age 35 y, smoker during pregnancy, pre-term birth < 37, pre-eclampsia, postpartum infection, postpartum hemorrhage, VTE family history).

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuelle LE MOIGNE, MD, PhD, Principal Investigator — CHU de Brest
Locations (18):
- France (18):
  - CHU d'Amiens Picardie, Amiens
  - CHU de Bordeaux, Groupe Pellegrin, Centre Aliénor d'Aquitaine, Bordeaux
  - CHU de Brest, Brest
  - Hôpital Béclère, AP-HP, Clamart
  - CHU de Clermont Ferrand Site Estaing, Clermont-Ferrand
  - CH départemental de Vendée, La Roche-sur-Yon
  - Hôpital Bicêtre, AP-HP, Le Kremlin-Bicêtre
  - Hôpital Nord Marseille, AP-HM, Marseille
  - Centre Hospitalier des Pays de Morlaix, Morlaix
  - CHRU de Nancy, Nancy
  - CHU de Nantes, Nantes
  - Hôpital Lariboisière, AP-HP, Paris
  - Groupe Hospitalier Paris Saint Joseph, Paris
  - CH de Pau, Pau
  - Centre Hospitalier de Périgueux, Périgueux
  - Centre Hospitalier de Cornouaille Quimper Concarneau, Quimper
  - CHU de Rennes, Rennes
  - CHU de St Etienne - Hôpital Nord, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning five years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.